CLINICAL TRIAL: NCT00965003
Title: High Resolution MRI in the Evaluation of Laryngeal Neoplasia
Brief Title: MRI Laryngeal Imaging With a Surface Coil
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Absence of key personnel to conduct study
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Edward J. Damrose, Associate Professor of Otolaryngology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ENT0019; 96536 (Other: Stanford University Alternate IRB Approval Number); SU-05292009-2661 (Other: Stanford University)
Record Dates: First submitted 2009-08-21; First posted 2009-08-25 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Laryngeal Neoplasms; Head and Neck Cancers; Larynx Cancer
MeSH Terms: conditions — Laryngeal Neoplasms; Head and Neck Neoplasms | interventions — Magnetic Resonance Spectroscopy; Postmortem Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MRI scan with surface coil (Experimental): Patients with known laryngeal cancer, with suspected cartilage involvement by conventional computed tomography scanning, who undergo high resolution magnetic resonance imaging enhanced with a surface coil placed over the larynx.
  Interventions: Procedure: MRI scan

INTERVENTIONS:
Procedure: MRI scan — Standard of Care
  Other Names: Magnetic Resonance Imaging; nuclear magnetic resonance imaging; magnetic resonance tomography

SUMMARY:
To determine if high resolution MRI can detect early invasion of cartilage by laryngeal carcinoma, and to determine if high resolution MRI may be superior to conventional MRI imaging or CT imaging to detect cartilage invasion.

DETAILED DESCRIPTION:
The purpose of this study is to use a new MRI imaging coil developed for enhancing structures made of cartilage to determine if the device can produce improved images of the human larynx. In addition, if enhanced images can be obtained, a further purpose will be to determine if, in patients with laryngeal cancer, whether or not early invasion of cartilage can be detected. Patients with laryngeal cancer will be asked to undergone an MRI scan using this new image-enhancing coil to see if cartilage invasion can be detected. Patients will be followed during and after treatment to determine their ultimate response to treatment. No additional MRI scans for the purposes of this protocol will be performed other than the initial pretreatment scan.

We hope to determine if this new MRI imaging device can detect early cancer invasion of the laryngeal cartilages in patients with laryngeal cancer. Since this modality has never been attempted before on the human larynx, we are simply looking for the presence or absence of cartilage destruction. Both conventional CT and conventional MRI are poor at recongnizing this finding. High resolution MRI may allow the detection of this finding or it may not - detection of this finding is the endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Patients with benign or malignant neoplasm of the larynx.
* Patients who have undergone prior surgery, radiation therapy, or chemotherapy for cancer of the laryngopharynx will be eligible to participate.
* Patients 18 years of age and older at time of evaluation, male and female, all ethnicities.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Pregnancy
* Claustrophobia.
* Anatomic parameters which preclude scanning, such as limited range of neck motion, or inability to remain flat for at least 15 minutes.
* Patients with implanted devices (eg, defibrillator, pacemaker) that are a known contraindication to magnetic resonance imaging.
* Allergy to gadolinium contrast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Tumor stage as determined by HRMRI. | 24 to 48 hours
  Radiologic tumor stage

SECONDARY OUTCOMES:
Estimate the precision of HRMRI in discriminating between edema and tumor in patients with prior radiotherapy or chemotherapy. | 4 to 6 weeks
  Comparison of true tumor dimension as predicted by HRMRI versus true tumor size as shown on final histopathology
Tumor stage as determined by histopathology in excised larynges. | 4 to 6 weeks
  Pathological tumor stage

CONTACTS AND LOCATIONS:
Overall Officials: Edward J. Damrose MD, FACS, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States